CLINICAL TRIAL: NCT06934421
Title: Segurança e eficácia de Nova Abordagem Ecoguiada de ablação Por radiofrequência Dos Nervos Geniculados
Brief Title: Revised Targets for Knee Radiofrequency Ablation
Acronym: ReTaKRA
Status: Recruiting | Type: Observational
Sponsor: Centro Hospitalar Universitario do Algarve (Other)
Responsible Party: Principal Investigator, Manuel Tomás Farinha Caroço, Medical Doctor, Centro Hospitalar Universitario do Algarve
Other Study IDs: 025/2025
Record Dates: First submitted 2025-04-10; First posted 2025-04-18 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Osteoarthritis Knee Pain
Keywords: Genicular nerve; Knee pain; Chronic pain; Knee osteoarthritis; Radiofrequency ablation; Ultrasound guidance; Interventional pain management; Joint degeneration; Nerve ablation; Image-guided procedures; Non-surgical treatment; Musculoskeletal intervention; Pain reduction; Functional improvement
MeSH Terms: conditions — Chronic Pain; Osteoarthritis, Knee | interventions — Radiofrequency Ablation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Single-Session Ultrasound-Guided Genicular Nerve Radiofrequency Ablation in Patients With Knee Osteo: Participants with knee osteoarthrosis (Kellgran-Lawrence III or IV) will receive a single-session ultrasound-guided radiofrequency ablation of the genicular nerves. The procedure targets three specific nerve branches around the knee joint: the superomedial, superolateral, and inferomedial genicular nerves. The targeted positions are based on anatomical reference points described by Fonkoue et al. (2021) and validated in cadaveric studies, aiming to improve the accuracy of nerve localization. Under ultrasound guidance, the clinician will insert a radiofrequency needle at each target site. After confirming correct positioning through sensory and motor stimulation, thermal ablation will be performed at 85ºC for 90 seconds per site. Local anesthesia will be administered before each ablation to ensure patient comfort. This procedure aims to reduce knee pain and improve function in patients with moderate to severe knee joint degeneration who have not responded to conservative treatments.
  Interventions: Device: Ultrasound-Guided Genicular Nerve Radiofrequency Ablation

INTERVENTIONS:
Device: Ultrasound-Guided Genicular Nerve Radiofrequency Ablation — This intervention involves a single-session ultrasound-guided thermal radiofrequency ablation of the superomedial, superolateral, and inferomedial genicular nerves in patients with moderate to severe knee osteoarthritis. Target points follow anatomical references described by Fonkoue et al. and validated in cadaveric studies, differing from classical approaches. Under ultrasound guidance, monopolar RF cannulas are placed, with sensory and motor stimulation confirming accurate positioning. Local anesthesia (2% lidocaine) is applied. Lesions are performed at 85°C for 90 seconds per site. The radiofrequency generator used is CE-marked for pain procedures. The study evaluates a novel targeting protocol, not the safety or effectiveness of the device itself. No fluoroscopy is used. The procedure is performed once. Participants are followed for two years to assess outcomes.
  Other Names: Thermal Radiofrequency Ablation of Genicular Nerves; Monopolar Radiofrequency Ablation of Knee Nerves; Image-Guided Genicular Nerve Ablation; Ultrasound-Guided RFA of Knee; Genicular Nerve RFA; RFA for Knee Osteoarthritis Pain

SUMMARY:
This research team is doing a study to learn more about a new way to treat long-term knee pain caused by joint damage. They are using a treatment called radiofrequency ablation (RFA). This is a procedure where doctors use heat to stop certain nerves from sending pain signals.

In this study, doctors will use ultrasound to guide a small needle to nerves around the knee, called genicular nerves. Then, they will apply heat to those nerves using radiofrequency energy to help reduce pain.

The team created this new method based on recent studies of knee anatomy. They want to find out if this method can safely reduce pain and help people with knee joint damage move better. The study includes people who have moderate to severe knee damage and still have pain after trying medicine, physical therapy, or joint injections.

Each person in the study will have the treatment once. The research team will follow each person for two years. During this time, people in the study will answer simple questions about their knee pain and how it affects their daily life. The researchers will collect this information before the treatment and several times after it. One week after the procedure, the team will call each person to ask how they are feeling and check for any side effects.

Possible benefits of the study include less knee pain and easier movement. Possible risks include pain during the procedure, bruising, swelling, or short-term worsening of pain. Rare risks include nerve problems, weakness, bone damage, or allergic reaction.

The study is free for participants, and there is no payment. Taking part is voluntary. Anyone can stop being in the study at any time without affecting their medical care. The research team will keep all personal information private and secure.

DETAILED DESCRIPTION:
This study applies a modified ultrasound-guided radiofrequency ablation (RFA) protocol for targeting the genicular nerves, informed by recent anatomical research. Conventional genicular nerve RFA techniques commonly rely on fluoroscopic or ultrasound guidance based on standard anatomical landmarks. However, cadaveric studies-such as those by Fonkoue et al. (2021)-have shown that these conventional approaches frequently miss the intended nerves, particularly the superomedial and superolateral branches, leading to inconsistent or suboptimal outcomes.

To address these limitations, this protocol incorporates revised probe positioning and alternative bony landmarks aligned with verified nerve pathways. The updated targeting strategy is designed to improve the precision and reproducibility of genicular nerve localization using high-resolution musculoskeletal ultrasound.

The procedure begins with ultrasound identification of the target genicular nerves. Once confirmed, a local anesthetic (2% lidocaine, 20-40 mg per site) is infiltrated to minimize discomfort. Thermal lesioning is then performed using standard 20G RF cannulas at 85°C for 90 seconds. Sensory stimulation (0.2-0.5 V) is used to verify appropriate referral patterns, and motor stimulation (2.0 V) is applied to rule out motor involvement before lesioning. If motor responses are elicited, repositioning or procedure cancellation is considered.

This anatomically informed technique aims to enhance procedural accuracy and consistency. By integrating cadaver-based nerve mapping with real-time ultrasound imaging, the approach has the potential to improve treatment effectiveness while maintaining a strong safety profile. The study will contribute clinical data supporting the feasibility and utility of this refined targeting method in managing knee pain related to joint degeneration.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic knee pain related to radiographic knee osteoarthritis, Kellgren-Lawrence (KL) grade III or IV, who are refractory to conservative treatment.

(Refractoriness to conservative treatment is defined as:

* Persistent pain and functional limitation after undergoing knee-targeted physiotherapy and analgesic medication in accordance with clinical guidelines for osteoarthritis [e.g., paracetamol, nonsteroidal anti-inflammatory drugs, and other drugs as deemed appropriate by the treating physician];
* Persistent pain and functional limitation after intra-articular corticosteroid injections or limited success with such interventions.)

Exclusion Criteria:

* Patients with previous knee arthroplasty
* Patients who have undergone prior radiofrequency (RF) ablation
* Significant psycho-emotional disorders
* Addictive behaviors
* Generalized pain
* Nociplastic pain
* Presence of a pacemaker
* Presence of osteosynthesis material in the knee or adjacent anatomical regions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from the community referred to the Physical and Rehabilitation Medicine department.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-03-20 (Actual); Primary Completion 2028-07-14 (Estimated); Study Completion 2031-07-30 (Estimated)

PRIMARY OUTCOMES:
Change in Knee Pain Intensity (Numeric Pain Rating Scale - NPRS) | Baseline to 3 months post-procedure
  Change in patient-reported knee pain at rest and during movement, measured using an 11-point Numeric Pain Rating Scale (0 = no pain, 10 = worst imaginable pain).

SECONDARY OUTCOMES:
Change in Physical Function (WOMAC Functional Subscale) | Baseline to 3 months, 6 months, 1 year, and 2 years post-procedure
  Change in physical function as measured by the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) - Physical Function Subscale. The WOMAC is a validated, self-reported questionnaire assessing functional limitations due to knee osteoarthritis.
  This subscale includes 17 items, each scored on a Likert scale from 0 to 4. The total score ranges from 0 to 68, with higher scores indicating worse physical function.
Sustained Pain Reduction (Numeric Pain Rating Scale) | Baseline to 1 week, 1 month, 3 months, 6 months, 1 year, and 2 years post-procedure
  Change in pain intensity over time as measured by the Numeric Pain Rating Scale (NPRS). The NPRS is an 11-point scale ranging from 0 to 10, where 0 represents "no pain" and 10 represents "worst imaginable pain". Patients will report their average knee pain intensity over the past 24 hours. Higher scores indicate worse pain. This outcome assesses the duration and consistency of the analgesic effect following the radiofrequency ablation procedure.
Incidence of Adverse Events | From procedure day to 2-year follow-up
  Number and type of adverse events related to the intervention, including local site pain, edema, bruising, motor weakness, neuritis, or other complications.
Responder Rate (≥50% Pain Reduction) | Baseline to 3 months post-procedure
  Proportion of participants achieving ≥50% reduction in NPRS at 3 months post-procedure compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Tomás Farinha Caroço, Medical Doctor, Principal Investigator — Unidade Local de Saude do Algarve / Centro Hospitalar Universitario Algarve
Locations (2):
- Portugal (2):
  - Serviço de Medicina Física e de Reabilitação - Hospital de Faro - Unidade Local de Saúde do Algarve, Faro
  - Serviço de Medicina Física e de Reabilitação - Hospital de São Francisco Xavier - Unidade Local de Saúde de Lisboa Ocidental, Lisbon

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that underlie the results reported in publications will be shared. This includes pain scores, functional outcomes (WOMAC), adverse event data, and baseline clinical and demographic variables such as age, sex, body mass index (BMI), radiographic knee imaging (image and Kellgren-Lawrence grade), painful knee quadrant, presence of depressive symptoms, and use of opioids, antidepressants, or anxiolytics. A data dictionary will be provided to support interpretation of the dataset.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Individual participant data (IPD) and supporting information will be available beginning 6 months after publication of the primary results. Data will remain available for a period of 5 years.
Access Criteria: Researchers who wish to access individual participant data (IPD) must submit a written request including a clear research question, rationale, and a detailed statistical analysis plan. The proposed analyses must be scientifically sound, ethically appropriate, and feasible given the dataset. Proposals must demonstrate consistency with the objectives of academic, non-commercial research.
  All requests will be reviewed by the principal investigator and the study's coordinating research team to ensure alignment with ethical standards and scientific merit. If the request is approved, the researcher will be required to sign a data sharing agreement that outlines the terms of use, including data confidentiality, appropriate use, and prohibition of re-identification.
  Approved data will be shared in de-identified format through a secure institutional repository or via encrypted file transfer. Requests and supporting documents can be submitted by email to the principal investigator.

REFERENCES:
- [Background] Cohen SP, Bhaskar A, Bhatia A, Buvanendran A, Deer T, Garg S, Hooten WM, Hurley RW, Kennedy DJ, McLean BC, Moon JY, Narouze S, Pangarkar S, Provenzano DA, Rauck R, Sitzman BT, Smuck M, van Zundert J, Vorenkamp K, Wallace MS, Zhao Z. Consensus practice guidelines on interventions for lumbar facet joint pain from a multispecialty, international working group. Reg Anesth Pain Med. 2020 Jun;45(6):424-467. doi: 10.1136/rapm-2019-101243. Epub 2020 Apr 3. PMID 32245841
- [Background] Pardal, Margarida Alexandra Rodrigues. Adaptação cultural para português europeu do Western Ontario and McMaster Universities Arthritis Index (WOMAC). Master's Thesis 2023;
- [Background] De Cassai A, Dost B, Tulgar S. Enhancing the clarity and reproducibility of regional anesthesia techniques: a call for video integration in scientific publications. Reg Anesth Pain Med. 2025 Oct 6;50(10):842-843. doi: 10.1136/rapm-2024-105871. No abstract available. PMID 39043621
- [Background] Tran J, Peng P, Agur A. Evaluation of nerve capture using classical landmarks for genicular nerve radiofrequency ablation: 3D cadaveric study. Reg Anesth Pain Med. 2020 Nov;45(11):898-906. doi: 10.1136/rapm-2020-101894. Epub 2020 Sep 14. PMID 32928998
- [Background] Tran J, Peng PWH, Chan VWS, Agur AMR. Overview of Innervation of Knee Joint. Phys Med Rehabil Clin N Am. 2021 Nov;32(4):767-778. doi: 10.1016/j.pmr.2021.05.011. Epub 2021 Jul 14. PMID 34593142
- [Background] Fonkoue L, Stoenoiu MS, Behets CW, Steyaert A, Kouassi JK, Detrembleur C, Cornu O. Validation of a new protocol for ultrasound-guided genicular nerve radiofrequency ablation with accurate anatomical targets: cadaveric study. Reg Anesth Pain Med. 2021 Mar;46(3):210-216. doi: 10.1136/rapm-2020-101936. Epub 2020 Dec 3. PMID 33273065
- [Background] Fonkoue L, Behets C, Kouassi JK, Coyette M, Detrembleur C, Thienpont E, Cornu O. Distribution of sensory nerves supplying the knee joint capsule and implications for genicular blockade and radiofrequency ablation: an anatomical study. Surg Radiol Anat. 2019 Dec;41(12):1461-1471. doi: 10.1007/s00276-019-02291-y. Epub 2019 Jul 23. PMID 31338537
- Available data/document: Study Protocol — https://osf.io/8ywq6/
- Available data/document: Statistical Analysis Plan — https://osf.io/8ywq6/
- Available data/document: Informed Consent Form — https://osf.io/8ywq6/
- Available data/document: Analytic Code — https://osf.io/8ywq6/
- Available data/document: Individual Participant Data Set — https://osf.io/8ywq6/